CLINICAL TRIAL: NCT03097601
Title: ELR+CXCL Cytokines in Metastatic Kidney Cancers: Predictive Markers of Resistance to Sunitinib and New Relevant Therapeutic Targets in Refractory Patients
Brief Title: ELR+CXCL Cytokines in Metastatic Kidney Cancers: Predictive Markers of Resistance to Sunitinib
Acronym: SUNITRES
Status: Completed | Type: Observational
Sponsor: Centre Antoine Lacassagne (Other)
Collaborators: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Other Study IDs: 2016/09
Record Dates: First submitted 2017-03-27; First posted 2017-03-31 (Actual); Last update posted 2020-07-21 (Actual); Status verified 2020-07

CONDITIONS: Metastatic Kidney Cancers
MeSH Terms: conditions — Kidney Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Experiment on cell lines, on human samples and animal models. CXCL cytokines as predictive markers of sunitinib efficacy in order to demonstrate the mechanisms linked to the production of CXCL cytokines by mRCC or in response to treatments
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- sunitinib cohort: independent cohorts of patients who received sunitinib for metastic kidney cancer, on who we intend to demonstrate that ELR+CXCL cytokines levels are of sunitinib response
  Interventions: Diagnostic Test: ELR+CXCL cytokines levels are of sunitinib response

INTERVENTIONS:
Diagnostic Test: ELR+CXCL cytokines levels are of sunitinib response — Demonstrate on independent cohorts of patients that ELR+CXCL cytokines levels are of sunitinib response

SUMMARY:
Metastatic renal cell carcinomas (mRCC) are highly angiogenic tumors because of mutation of the pVHL gene leading to over-expression of VEGF. Therefore, mRCC represent a paradigm for the use of anti-angiogenic treatments targeting the VEGF/VEGFR pathway. Despite an increase of the time to progression these treatments, taken alone, are not curative with ineluctable progression especially for the reference treatment sunitinib a multi kinase inhibitors of VEGF, PDGF, CSF1 receptors and c-kit, FLT3 and RET. At progression on sunitinib, patients received mTOR inhibitors which is responsible, at least, of HIF1A mRNA translation, then on a third line sorafenib that inhibits VEGFR2, 3 PDGFR, c-KIT and B-RAF. The access to these different lines of treatment has finally prolonged survival but this situation is not satisfactory. Unexpected aspect associated with the use of anti-angiogenesis treatments was the diversity of the patients' response. Some patients are right away refractory and die rapidly, but the majority of patient has a transient response then progress and a few percentages of them are responder for a very long period of time. By only targeting normal endothelial cells and tumor neo-vascularization, the response should have been more homogenous, thus highlighting that the treatment induced a "Darwinian" adaptation of tumor cells and cells of the microenvironment. Two conclusions follow from these observations: 1- The need to identify predictive markers of efficacy; 2-The identification of druggable targets participating in progression on anti-angiogenic treatments. Our results have highlighted the ELR+CXCL cytokines, pro-inflammatory and pro-angiogenic cytokines as prognosis markers of survival of mRCC patients and relevant therapeutic targets on experimental tumors in mice. As VEGF/VEGFR, these cytokines are produced by tumor, endothelial and inflammatory cells. Their receptors (CXCR1, 2) are expressed physiologically by immune and endothelial cells and aberrantly by tumor cells generating at the same time autocrine proliferation loops, chronic angiogenesis and inflammation. Therefore, the CXCL/CXCR1,2 axis constitutes an independent axis of cancer development and propagation. However, the current standard of care is to administer anti-angiogenic therapies as the first line treatment. The objective of this project is linked to the identification of potent predictive markers of efficacy, easily measured in plasma samples. Deciphering the molecular mechanisms associated with the production of such cytokines by tumor cells and by cells of the microenvironment represents an interesting intellectual challenge and a relevant way to improve the current treatments by targeting, at progression on the current standard of care, other pathways than the VEGF/VEGFR axis.

DETAILED DESCRIPTION:
Metastatic renal cell carcinomas (mRCC) are highly angiogenic tumors because of mutation of the pVHL gene leading to over-expression of VEGF. Therefore, mRCC represents a paradigm for the use of anti-angiogenic treatments targeting the VEGF/VEGFR pathway. Despite an increase of the time to progression these treatments, administered alone, are not curative with ineluctable progression especially for the reference treatment sunitinib a multi kinase inhibitors of VEGF, PDGF, CSF1 receptors and c-kit, FLT3. At progression with sunitinib treatment, patients received mTOR inhibitors which is responsible, at least, of HIF1A mRNA translation, then through a third line sorafenib that inhibits VEGFR2, 3 PDGFR, c-KIT and B-RAF. The access to these different lines of treatment has finally prolonged survival but this situation is not satisfactory. New way of thinking and new therapeutic targets are necessary to "chronisize" the pathology or even to cure it. The current therapeutic practises are based on the statement that the treatments must destroy blood vessels to asphyxiate the tumors and that endothelial cells are normal cells that cannot adapt to the selection pressure exerted by the treatments. These statements arewrong since tumor cells aberrantly express the receptors targeted by anti-angiogenic drugs leading to cell adaptation and tumor recurrence. Another unexpected aspect associated with the use of anti-angiogenesis treatments was the diversity of the patients'response. Some patients are right away refractory and die rapidly, but the majority of patients has a transient response then progress and a few percentages of them are responders for a very long period. By only targeting normal endothelial cells and tumor neo-vascularization, the response should have been more homogenous. 3 conclusions follow from these observations: 1- The need to identify predictive markers of efficacy; 2-The identification of druggable targets participating in progression on anti-angiogenic treatments; 3- These targets should be independent of the VEGF/VEGFR axis.

The results have highlighted the ELR+CXCL cytokines, pro-inflammatory and pro-angiogenic cytokines as prognosis markers of survival of mRCC patients and relevant therapeutic targets on experimental tumors in mice. As VEGF/VEGFR, these cytokines are produced by tumor, endothelial and inflammatory cells. Their receptors (CXCR1, 2) are expressed physiologically by immune and endothelial cells and aberrantly by tumor cells generating at the same time autocrine proliferation loops, chronic angiogenesis and inflammation. Therefore, the CXCL/CXCR1,2 axis constitutes an independent axis of cancer development and propagation. However, the current standard of care is to administer anti-angiogenic therapies as the first line treatment. Hence, what is the relevance of CXCL cytokines as predictive markers of sunitinib efficacy, and what are the mechanisms linked to the production of CXCL cytokines by mRCC or in response to treatments?. Deciphering the molecular mechanisms associated with the production of such cytokines by tumor cells and by cells of the microenvironment represents an interesting intellectual challenge and a relevant way to improve the current treatments by targeting, at progression on the current standard of care, other pathways than the VEGF/VEGFR axis.

This project aimed at the improvement of current clinical practises for mRCC. Numerous efforts have been given to the determination of prognosis markers for different tumors including mRCC. However, for clinical practises, physicians are more interested to predictive markers of success/failure of a treatment that to biological prognosis markers that are most of the time as indicative as classical clinical parameters (TNM for example). The recent experiments have highlighted relevant cytokines (ELR+CXCL) participating in the aggressiveness of mRCC. Indeed, the intra-tumor amounts of the ELR+CXCL cytokine CXCL7 was a potent prognosis marker of survival independent of any clinical parameters. Therefore it was indicative of poor prognosis for patients who were a priori of good prognosis according to the TNM or the Fuhrman grade (consideration of nuclear and nucleolus size). We have also demonstrated the prognosis value of two other ELR+CXCL cytokine CXCL1, CXCL5 and CXCL8. Both of them are not independent of clinical parameters. However, their role as predictive markers of resistance to anti-angiogenic drugs, the current standard of care, is still unknown.

For a medical point of view, a rapid identification of responders and no-responders is of first importance. It will avoid undesired toxic events for unresponsive patients and a rapid adaptation of the treatment considering that different lines of therapies are currently available for mRCC patients. The determination of a threshold value for the most relevant cytokines is needed and this threshold must be determined of independent cohort of patients for a better reliability. Such test should not be invasive for the patients and as simple as possible in order to introduce in clinical practises for a low price that can be reimburse by the social security. It is compatible with what we propose to do by measuring ELR+CXCL levels on blood samples with classical ELISA tests.

Deciphering the mechanisms at the origin of the de novo synthesis of redundant pro-angiogenic/pro-inflammatory cytokines under the selection pressure of treatment targeting the VEGF/VEGFR pathway is intellectually challenging and may identify unknown parameters implicated in Darwinian adaptation of tumor cells among a very heterogeneous environment.

The main objectives are :

* Research helping to the understanding of biological mechanisms from clinical observations (Bed to Bench) and the transfer of knowledge from the clinic to the laboratories (bed to bench).
* Research helping to the prognosis.
* Research helping to the therapeutic decision and treatment monitoring.

ELIGIBILITY:
Inclusion Criteria:

* patients with mRCC and treated by sunitinib after radical nephrectomy included in SUVEGIL 8 Clinical Trial (Sponsor : Centre Antoine Lacassagne)

Exclusion Criteria:

* Non applicable

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with mRCC and treated by sunitinib after radical nephrectomy
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2016-06-02 (Actual); Primary Completion 2019-12-30 (Actual); Study Completion 2019-12-30 (Actual)

PRIMARY OUTCOMES:
ELR+CXCL cytokines | December 2018
  To determine of a threshold level of one or multiple ELR+CXCL cytokines indicative of progression for routine clinical practises

SECONDARY OUTCOMES:
molecular mechanisms | December 2020
  To decipher the molecular mechanisms implicated in ELR+CXCL cytokines expression at the basal level and at progression on sunitinib. Expression of these cytokines by tumor cells and cells from the microenvironment (especially the Macrophages M1/Macrophages M2 ratio).

CONTACTS AND LOCATIONS:
Overall Officials: Christine LOVERA, Study Director — Centre Antoine Lacassagne
Locations (1):
- Centre Antoine LACASSAGNE, Nice, France

IPD SHARING:
Plan to Share IPD: No